CLINICAL TRIAL: NCT01251055
Title: GlyT-1 Inhibitor Treatment for Refractory Schizophrenia and Its Effects on NMDA Modulation
Brief Title: GlyT-1 Inhibitor Treatment for Refractory Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Hsien-Yuan Lane, Department of Psychiatry, China Medical University Hospital, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMR-98-096
Record Dates: First submitted 2010-11-03; First posted 2010-12-01 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Schizophrenia; Treatment Refractory
Keywords: N-methyl-D-aspartate receptor; glycine transporter; schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- GlyT-1 inhibitor-1 (Experimental): GlyT-1 inhibitor-1 4000 mg/day
  Interventions: Drug: GlyT-1 inhibitor-1

INTERVENTIONS:
Drug: GlyT-1 inhibitor-1 — GlyT-1 inhibitor-1(500) 4# BID
  Arms: GlyT-1 inhibitor-1
Drug: Placebo — starch
  Arms: Placebo

SUMMARY:
The etiology of schizophrenia remains unclear In recent one decade, hypofunction of N-methyl-D-aspartate (NMDA) receptor has been implicated in the pathophysiology of schizophrenia. Hence, enhancing NMDA neurotransmission was considered as a new approach for schizophrenia treatment.

To date, refractory schizophrenia (particularly clozapine-resistant) is still a difficult clinical issue. However, the effect of NMDA treatment in refractory schizophrenia is still unknown. Therefore, the primary goal of this study is to investigate the efficacy and safety of NMDA adjuvant therapy in refractory schizophrenia, and to identify the predictors for treatment response to NMDA enhancers.

DETAILED DESCRIPTION:
The etiology of schizophrenia remains unclear. In recent one decade, hypofunction of N-methyl-D-aspartate (NMDA) receptor has been implicated in the pathophysiology of schizophrenia. Hence, enhancing NMDA neurotransmission was considered as a new approach for schizophrenia treatment. To date, there have been a few pilot studies exploring the efficacy of NMDA enhancers as adjuvant therapy for schizophrenia, for instance, D-serine (an endogenous agonist of the NMDA-glycine site). They were not only well-tolerated but also synergistic in improving positive, negative and cognitive symptoms in those receiving typical and atypical antipsychotics (except clozapine).

Refractory schizophrenia (particularly clozapine-resistant) is still a difficult clinical issue at present. Previous studies revealed that add-on treatment of D-serine or other agonists of NMDA receptor failed to give significant benefits in such patients. The primary goal of this study is to investigate the efficacy and safety of glycine transporter(GlyT)-1 inhibitor adjuvant therapy in refractory schizophrenia, and to identify the predictors for treatment response to NMDA enhancers.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill the criteria of schizophrenia according to the Diagnostic and Statistic Manual, fourth edition (DSM-IV).
* Poor response of clozapine treatment: a 12-week treatment of clozapine without satisfactory response: a severity score of Clinical Global Impression Scale(CGI)>=4, a total score of Positive and Negative Syndrome Scale(PANSS)>= 60, and a Scale for the Assessment of Negative Symptoms(SANS)score of >=40. the doses of clozapine remain stable for at least 12 weeks prior to their enrollment in this proposed study,
* Agree to participate in the study and provide informed consent.

Exclusion Criteria:

* current substance abuse or history of substance dependence in the past 6 months
* use of depot antipsychotic in the past 6 months
* serious medical or neurological illness
* pregnancy
* inability to follow protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The severity of psychiatric symptoms | baseline
  The severity of psychiatric symptoms will be assessed by:
  1. Positive and Negative Syndrome Scale(PANSS)
  2. Assessment of Negative symptoms(SANS)
  3. Global assessment of function(GAF)
The severity of psychiatric symptoms | 2 weeks after the trial
  The severity of psychiatric symptoms will be assessed by:
  1. Positive and Negative Syndrome Scale(PANSS)
  2. Assessment of Negative symptoms(SANS)
  3. Global assessment of function(GAF)
The severity of psychiatric symptoms | 4 weeks after the trial
  The severity of psychiatric symptoms will be assessed by:
  1. Positive and Negative Syndrome Scale(PANSS)
  2. Assessment of Negative symptoms(SANS)
  3. Global assessment of function(GAF)
The severity of psychiatric symptoms | 6 weeks after the trial (The end of the trial)
  The severity of psychiatric symptoms will be assessed by:
  1. Positive and Negative Syndrome Scale(PANSS)
  2. Assessment of Negative symptoms(SANS)
  3. Global assessment of function(GAF)

SECONDARY OUTCOMES:
Neurocognitive Function | baseline
  The neurocognitive functions will be assessed by:
  1. Wisconsin Card Sorting Test (WCST)
  2. Wechsler Memory Scale- logical memory
Neurocognitive function | 6 weeks after the trial (The end of the trial)
  The neurocognitive functions will be assessed by:
  1. Wisconsin Card Sorting Test (WCST)
  2. Wechsler Memory Scale- logical memory
The severity of psychiatric symptoms | baseline
  The severity of psychiatric symptoms will be assessed by:
  1. Clinical Global Impression(CGI)
  2. Subscales of PANSS
The severity of psychiatric symptoms | 2 weeks after the trial
  The severity of psychiatric symptoms will be assessed by:
  1. Clinical Global Impression(CGI)
  2. Subscales of PANSS
The severity of psychiatric symptoms | 4 weeks after the trial
  The severity of psychiatric symptoms will be assessed by:
  1. Clinical Global Impression(CGI)
  2. Subscales of PANSS
The severity of psychiatric symptoms | 6 weeks after the trial (the end of the trial)
  The severity of psychiatric symptoms will be assessed by:
  1. Clinical Global Impression(CGI)
  2. Subscales of PANSS

CONTACTS AND LOCATIONS:
Overall Officials: Hsien-Yuan Lane, MD.PhD., Principal Investigator — Department of Psychiatry, China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan, Taiwan